CLINICAL TRIAL: NCT02433028
Title: Swiss Multiple Sclerosis Cohort-Study: A Prospective Swiss Wide Investigation of Key Phases in Disease Evolution and New Treatment Options
Brief Title: Swiss Multiple Sclerosis Cohort-Study
Acronym: SMSC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Cantonal Hospital of Aarau, Switzerland (Other); Cantonal Hospital of St. Gallen (Other); Insel Gruppe AG, University Hospital Bern (Other); Regional Hospital Lugano (EOC), Switzerland (Unknown); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other); National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Other Study IDs: SMSC_1_3
Record Dates: First submitted 2014-12-18; First posted 2015-05-04 (Estimated); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: MS key phases of disease evolution; MS New Treatment Options
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Swiss MS Cohort Study (SMSC) is a multicentre cohort study that involves 8 Swiss Multiple Sclerosis centres. The key aims of the SMSC are

1. To maintain a long-term cohort for an undefined duration of patients with Multiple Sclerosis (MS), neuromyelitis optica spectrum disorder (NMOSD) and Myelin oligodendrocyte glycoprotein antibody-associated disease (MOGAD) in Switzerland. This requires effective measures to limit drop-outs and the continuous recruitment of MS patients and
2. To conduct a systematic follow-up with standardized, high quality collection of clinical and magnetic resonance imaging (MRI) data, as well as body fluids.

The significant heterogeneity within the diagnostic entity and phenotype of MS is incompletely understood. A central and necessary prerequisite of further advance is a sufficient amount of high quality clinical and paraclinical (imaging, body fluids) patient data.

Nested projects will address specific research topics, and facilitate collaboration of the most qualified investigators within the group of SMSC investigators. The nested projects will focus on the:

1. Development and validation of diagnostic and prognostic markers of spontaneous disease evolution and therapeutic response.
2. Exploration of the safety and impact on long-term disability of existing and next generation MS treatments
3. Individualized therapy: A number of highly active but potentially also harmful therapies have lately been established for the treatment of MS. To date, due to the lack of individual prognostic markers patients may not receive aggressive therapy due to safety concerns, or patients with benign disease may receive expensive and potentially harmful treatments without the need for it.
4. Evaluation of intervention effects by conducting embedded pragmatic trials using the SMSC as data-infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the diagnosis of radiologically isolated syndrome (RIS), clinically isolated syndrome (CIS), relapsing-remitting Multiple Sclerosis (RRMS), secondary-progressive MS (SPMS), primary-progressive MS (PPMS), neuromyelitis optica spectrum disorder (NMOSD) or Myelin oligodendrocyte glycoprotein antibody-associated disease (MOGAD) according to established criteria
* Intending to attend hospital visits every 6 months (+/- 45 days) or 12 months (+/- 45 days) (facultative cranial MRI every 12 months) over a longer period (at least 5 years)
* Intending to give blood for biobanking every 6 or 12 months during hospital visit or as close as possible to the visit (+/- 8 days)

Inclusion criteria are crafted to identify a population of patients with MS, NMOSD or MOGAD particularly suitable for analysing disease evolution and associated factors, treatment dynamics, and the long-term safety and efficacy profile of disease-modifying drugs.

There are no specific Exclusion Criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of radiologically isolated syndrome (RIS), clinically isolated syndrome (CIS), relapsing-remitting MS (RRMS), secondary-progressive MS (SPMS), primary-progressive MS (PPMS), neuromyelitis optica spectrum disorder (NMOSD) or Myelin oligodendrocyte glycoprotein antibody-associated disease (MOGAD)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2042-01 (Estimated); Study Completion 2042-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Expanded Disability Status Scale (EDSS) | Baseline and at each follow-up visit (every 6 or 12 months)
  Expanded Disability Status Scale (EDSS) is measured using Neurostatus by certified neurologists
Assessment of the quality of life | Baseline and at least once a year
  To assess the quality of life, the following patient-reported outcomes are collected:
  * Multiple Sclerosis Quality of Life-54: A self-report questionnaire regarding quality of life with 36 generic (which corresponds to the 36 items of the Short-Form-36 questionnaire) and 18 MS-specific items.
  * EuroQoL-5D: A self-report questionnaire on generic quality of life, with one question for each of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). It also includes a Visual Analog Scale regarding perceived health status, ranging from 0 (worst possible) to 100 (best possible).
  * Patient reported questionnaire: Includes questions regarding professional activity and changes, and hospitalization.
Collection of serum and plasma (and, optional) cerebrospinal fluid samples | Baseline and at each follow-up visit (every 6 or 12 months)
  Serum and plasma samples will be collected every 6 or 12 months for all participants during study visit. Cerebrospinal fluid samples are facultative and contribute only if the participant is undergoing a diagnostic lumbar puncture.
(Optional) Assessment of finger dexterity | Baseline and at each follow-up visit (every 6 or 12 months)
  To assess the finger dexterity, the 9-Hole Peg Test is performed. It evaluates manual dexterity by measuring the time it takes for the participant to move nine pegs from a box into nine holes on a board and back. The 9-Hole Peg Test is not mandatory and is performed at the discretion of the physician.
(Optional) Electrophysiological assessment | Baseline and at each follow-up visit (every 6 or 12 months)
  To measure the visual, sensory and motor conduction time in the CNS, evoked potential tests are performed. Evoked Potentials are not mandatory and is performed at the discretion of the physician.
(Optional) Laboratory tests | Baseline and at each follow-up visit (every 6 or 12 months)
  The following laboratory tests are not mandatory, but are routinely performed in patients with MS at the discretion of the physician: Anti-JCV antibody test
  * Anti-natalizumab antibody test
  * Lymphocyte count
(Optional) Magnetic resonance imaging | Baseline and at least once per year
  The MRI is optional. All MRIs are collected that are done in clinical routine and follow the SMSC MRI protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kuhle, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (8):
- Switzerland (8):
  - Cantonal Hospital Aarau, Aarau, Canton of Aargau
  - University Hospital Basel, Basel, Canton of Basel-City
  - University Hospital Berne, Bern, Canton of Bern
  - University Hospital Geneva, Geneva, Canton of Geneva
  - Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Lausanne, Lausanne, Canton of Vaud
  - Regional Hospital Lugano, Lugano, Canton Ticino
  - Univeristy Hospital Zürich, Zurich